CLINICAL TRIAL: NCT05462119
Title: A Multicenter, Prospective, Non-interventional Cohort Study to Evaluate the Safety of Oral Resin for Treatment of Hyperkalemia in Chinese Patients With Renal Insufficiency
Brief Title: Safety of Oral Resin for Treatment of Hyperkalemia in Chinese Patients With Renal Insufficiency
Acronym: SCRUTINIZE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9483R00002
Record Dates: First submitted 2022-05-23; First posted 2022-07-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Hyperkalaemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a multicenter, prospective, non-interventional cohort study, in order to evaluate the safety of oral resin for treatment of hyperkalemia in Chinese patients with renal insufficiency.

DETAILED DESCRIPTION:
Background/Rationale:

Hyperkalaemia (HK) is a common electrolyte disturbance in clinical practice, defined as serum potassium (sK) beyond the normal range. The cut-off value for HK diagnosis is 5.0 mmol/L in most international guidelines[1, 2]. HK changes potassium ion gradient across the cell membrane and affects the excitability and conductivity of cardiomyocytes, leading to various types of arrhythmias, including ventricular arrhythmia, cardiac arrest and sudden death[3]. In the general population, the prevalence of HK is about 2-3%[4-6]. In an epidemiological survey in China, 3.86% of general outpatients experienced HK, and the proportion of patients who experienced HK increased in patients with chronic kidney disease (CKD), heart failure, diabetes and hypertension [7]. Furthermore，62% hospitalized HK patients accompanied by acute kidney injury (AKI)[8].

Treatment options for HK are well documented, and urgent therapy is indicated for rapid and substantial elevations in sK. However, for patients with modest elevations in sK without cardiac and neuromuscular manifestations, oral resin is in line with clinical practice, both calcium polystyrene sulphonate (CPS) and sodium polystyrene sulfonate (SPS), are applicable to HK caused by acute and chronic renal dysfunction.

CPS/SPS entraps potassium in the distal colon in exchange for calcium/ sodium to potassium. CPS may have an advantage over SPS because it avoids sodium retention. However, few clinical studies have evaluated the safety and efficacy of CPS/SPS in the treatment of HK. This study is expected to enhance and supplement the currently available CPS/SPS safety and effectiveness data in Chinese population in real world practice.

Objectives:

Primary objectives: To describe the safety and tolerability of CPS/SPS for HK management in Chinese patients with renal insufficiency in terms of adverse events (AEs), serious adverse events (SAEs) and discontinuations of CPS/SPS due to adverse events (DAEs).

Secondary objectives:

* To describe the safety and tolerability of CPS/SPS for HK management in Chinese hyperkalaemic patients with renal insufficiency in terms of AEs, SAEs and DAEs judged by the study investigators to be causally related to CPS/SPS.
* To understand the treatment pattern of CPS/SPS in real-world clinical practice for treating HK in Chinese patients with renal insufficiency.
* To describe the sK level of patients with renal insufficiency treated with CPS/SPS during the observational period

Methods:

Study design: The study is a multi-center prospective observational cohort study which will enroll patients who are ongoing and new users for HK management on CPS/SPS at study enrolment in real-world clinical practice. The eligible patients will be identified by physicians in each study site by assessing the patients or reviewing the medical record.

The prescription (including initiation, dose-adjusting or interruption) or discontinuation of CPS/SPS will be determined by physicians as per real-world clinical practice and in accordance with the local label. Any AstraZeneca (AZ) employee, or member of the research operation team will not intervene the decision-making of any physician or patient through any approach, at any time during the study.

Every patient will be followed up according to standard clinical practice for 6 months from enrolment.

At Study Enrolment Day (Day 1) the patients will be classified into 2 groups as new user group and ongoing user group. New users are defined that the patients starting CPS/SPS but without CPS/SPS treatment within 7 days before Day 1. Ongoing users are defined that the patients with CPS/SPS treatment within 7 days before Day 1 and continue CPS/SPS treatment after enrolment. The patients with previous CPS/SPS treatment who will not continue taking CPS/SPS treatment after enrolment will not be included.

Per standard clinical practice, new users of CPS/SPS should visit doctors within 1-3 days after initiation of treatment for potassium re-testing, then new users and ongoing users should visit doctors at Month 1, Month 3 and Month 6 for potassium monitoring or chronic disease consultation.

For new user group

* The "study index CPS/SPS treatment episode" starts at Study Enrolment Day.
* Follow-up visits will be planned on the 3rd day, the 1st month, the 3rd month and the 6th month from Study Enrolment Day.

For ongoing user group

* The "study index CPS/SPS treatment episode" started prior Study Enrolment Day.
* Follow-up visits will be planned on the 1st month, the 3rd month and the 6th month from Study Enrolment Day.

Visits of Day 1 (Study Enrolment Day) and Day 3 (only applicable for patients in new user group) are onsite. For visits at Month 1, Month 3 and Month 6, if the patient continues taking CPS/SPS treatment at the visit time points, the visit will be onsite. Otherwise, the visit will be conducted by phone-call. At each visit, safety outcomes, sK measurements data (if available), treatment data of CPS/SPS (as applicable) and other related data (if available) will be collected, as detailed in Section 6.1.2.

Data Source: This study will be based on primary (prospective) data collected from approximately 30 hospitals in China recruiting around 1000 patients. The site investigators will be responsible for ensuring that all the required data are collected and entered into the electronic case report form (eCRF).

Study Population: This study will enroll Chinese patients with renal insufficiency who are new users or ongoing users of CPS/SPS defined above at Study Enrolment Day. Eligible patients can be those with or without hemodialysis treatment.

Exposure: Treatment dose and duration of CPS/SPS is at the discretion of the patient's treating physician.

Outcome (s): Study measures will be collected at Day 1 and at the scheduled study visits.

Primary Endpoints:

• Occurrence of AEs, SAEs and DAEs during the study.

Secondary Endpoints:

* Occurrence of AEs, SAEs and DAEs judged by the investigators to be causally related to CPS/SPS.
* Average CPS/SPS daily dosage, frequency of different CPS/SPS dosages, duration of CPS/SPS treatment, dose changes and reasons for any dose changes.
* Change in sK tested between V1 and V2 (patients in new user group), as well as average (within patient) sK levels during the study. An evaluation of whether or not a patient tends to be normokalemic. Two criteria for normokalemia will be considered:

  * sK between 3.5 to 5.0 mmol/L, inclusive
  * sK between 3.5 to 5.5 mmol/L, inclusive. Sample Size Justification: Assuming the expected ratio of patients on SPS vs. CPS would be around 2:1, then with the total of 1,000 patients, the number of patients on SPS and CPS would be approximately 650 and 350.

Among 350 patients on CPS, new users and ongoing users are expected to be 150 and 200; While among 650 patients on SPS, new users and ongoing users are expected to be 300 and 350 Assuming the AE rate for different types of AE would be ranging from 1% to 12.8% for CPS [9]and 10% to 46.7% for SPS[10], current sample size could provide regarding 95% confidence interval (CI) as [0.1%, 5.7%] to [8.2%, 17.4%] for CPS and [6.6%, 13.4%] to [41.2%, 51.9%] for SPS, estimated using Normal Approximation and Clopper-Pearson's exact method (for AE rate of 1% only), which meets with general clinical requirements.

Sample size estimation under other scenarios as well as detailed description of estimation approach will be provided in section 5.4.

Statistical Analysis:

This study is primarily of descriptive character with no formal hypothesis testing for the objectives. The analyses will, as a rule, consist of estimates (of probabilities, rates, means, etc.), with the corresponding 95% CIs, as well as supportive descriptive statistics such as mean, standard deviation (SD), median, minimum, maximum, and quartiles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year-old
* Provision of patient informed consent prior to any study procedure
* Patients diagnosed as CKD or AKI
* HK (sK+ > 5.0 mmol/L) diagnosed by physicians within 1 year before Day 1
* Currently taking CPS/SPS, or have been prescribed and agree to start taking CPS/SPS since Day 1.

Exclusion Criteria:

* Being unable to comply with study-specified procedures
* Has ever participated in current study before, or participating in any interventional study at Day 1 or within the last 3 months before Day 1.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll eligible Chinese patients who are new and ongoing users on CPS/SPS at Study Enrollment from approximately 30 sites in China recruiting 1000 patients. New users are defined that the patients without CPS/SPS treatment within 7 days before Study Enrollment Day takeCPS/SPS treatment on Study Enrollment Day. Ongoing users are defined that the patients with CPS/SPS treatment within 7 days before Study Enrollment Day continue CPS/SPS treatment after enrollment. The patients with previous CPS/SPS treatment who will not continue taking CPS/SPStreatment after enrollment will not be included. Eligible patients will be those who meet all inclusion criteria but not any exclusion criteria. Eligible patients can be patients with or without hemodialysis treatment.
Sampling Method: Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of AEs | From enrollment to the 6th month after enrollment
  Number and percentage of AEs
Occurrence of SAEs | From enrollment to the 6th month after enrollment
  Number and percentage of SAEs
Occurrence of DAEs | From enrollment to the 6th month after enrollment
  Number and percentage of DAEs

SECONDARY OUTCOMES:
Occurrence of AEs judged by the investigators to be causally related to CPS/SPS | From enrollment to the 6th month after Enrollment
  Number and percentage of AEs judged by the investigators to be causally related to CPS/SPS
Occurrence of SAEs judged by the investigators to be causally related to CPS/SPS | From enrollment to the 6th month after Enrollment
  Number and percentage of SAEs judged by the investigators to be causally related to CPS/SPS
Occurrence of DAEs judged by the investigators to be causally related to CPS/SPS | From enrollment to the 6th month after Enrollment
  Number and percentage of DAEs judged by the investigators to be causally related to CPS/SPS
Average CPS/SPS daily dosage | From enrollment to the 6th month after enrollment
  Average CPS/SPS daily dosage
Frequency of different CPS/SPS dosages | From enrollment to the 6th month after enrollment
  Frequency of different CPS/SPS dosages
Duration of CPS/SPS treatment | From enrollment to the 6th month after enrollment
  Duration of CPS/SPS treatment
CPS/SPS dose changes | From enrollment to the 6th month after enrollment
  CPS/SPS dose changes
Reasons for any CPS/SPS dose changes | From enrollment to the 6th month after enrollment
  Reasons for any CPS/SPS dose changes
Change in sK tested between V1 and V2 (patients in new user group), as well as average (within patient) sK levels | From enrollment to the 6th month after enrollment
  Change in sK tested between V1 and V2 (patients in new user group), as well as average (within patient) sK levels during the study. An evaluation of whether or not a patient tends to be normokalemic. Two criteria for normokalemia will be considered:
  1. sK between 3.5 to 5.0 mmol/L, inclusive
  2. sK between 3.5 to 5.5 mmol/L, inclusive.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, Study Chair — Peking University People's Hospital
Locations (16):
- China (16):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Research Site, Beijing
  - Research Site, Dalian
  - Research Site, Dongyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kaifeng
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhangjiagang
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D9483R00002_Redacted_CSR synopsis. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9483R00002&attachmentIdentifier=d6e994c2-e670-41f1-a2eb-f8bfce15532e&fileName=D9483R00002_Redacted_CSR_synopsis.pdf&versionIdentifier=